CLINICAL TRIAL: NCT01665118
Title: The Cutera Trusculpt Device For Thigh Circumference Reduction
Brief Title: The Trusculpt (Radio Frequency) Device For Thigh Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-12-TS05
Record Dates: First submitted 2012-08-10; First posted 2012-08-15 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Body Fat
Keywords: Radio frequency; thigh; circumference; reduction

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (2):
- Treated Thigh (Experimental): Trusculpt (Radio Frequency) Device
  Interventions: Device: Trusculpt (Radio Frequency) Device
- Untreated Contra-lateral Thigh (No Intervention): To be used as the self control in this split body study.

INTERVENTIONS:
Device: Trusculpt (Radio Frequency) Device
  Arms: Treated Thigh

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the Trusculpt (Radio Frequency) device in the reduction of thigh circumference.

DETAILED DESCRIPTION:
The primary efficacy variable for this study is the comparison of mean change in thigh circumference from baseline to 12 weeks between two arms. The primary research hypothesis is that the mean change in thigh circumference is ≥ 1 cm (indicating mean reduction).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Minimum age of 18 years
* Non-smoking for at least 3 months and willing to refrain from smoking for the duration of the study.
* Post-menopausal, or on birth control and/or no plans to become pregnant for the duration of the study.
* Body Mass Index (BMI) ≤ 30
* Visible fat in the thigh / saddlebag area to be treated
* Subject must be able to read, understand and sign the Consent Form
* Subject must adhere to the follow-up schedule and study instructions
* Subject must adhere to the same diet and/or exercise routine throughout the study, and agree to maintain the same weight throughout the study (within 6 lbs of the weight measure at the baseline assessment)

Exclusion Criteria:

* Taking weight-loss medications/supplements
* Simultaneous participation in any other clinical study
* Prior surgical treatment to the target area, e.g., liposuction or abdominoplasty
* Prior treatment to the target area within the last 12 months e.g., radio frequency or cryolysis
* Arteriosclerosis or weakened blood vessels
* Heart disease
* Thromboembolic disease
* Diagnosed or documented immune system disorders (including Panniculitis)
* Bleeding disorders
* Presence of uncontrolled hypertension
* Taking prescription anticoagulants
* History of keloid formation
* History of malignant tumors in the target area
* Diabetes
* Any disease or condition that could impair wound healing
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles
* Infection in the target area
* Implanted electrical device(s) or metallic implants
* Pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Biesman, MD, Principal Investigator; Barry DiBernardo, MD, Principal Investigator; Stephen Ronan, MD, Principal Investigator
Locations (3):
- United States (3):
  - Cutera Research Center, Brisbane, California
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Nashville Center for Laser and Facial Surgery, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Thighs
Groups:
- All Study Participants: Subjects received RF treatments on one upper thigh (lateral and/or frontal and/or medial and/or posterior sides) according to randomization assignment and the opposite thigh served as the control.
Period: Overall Study
Arm/Group | All Study Participants
Started | 44; 88 Thighs
Thigh Treated With RF | 44; 44 Thighs
Untreated Thigh | 44; 44 Thighs
Completed | 26; 52 Thighs
Not Completed | 18; 36 Thighs

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: Subjects received RF treatments on one upper thigh (lateral and/or frontal and/or medial and/or posterior sides) according to randomization assignment and the opposite thigh served as the control.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Change of Thigh Circumference From Baseline
Description: Change in thigh circumference from baseline of the treated thigh compared to the non-treated contra-lateral side at 12 weeks post-final treatment.
Time Frame: Comparison of Baseline to 12 weeks post- final treatment
Measure: Mean (Full Range); unit: cm
Groups:
- Treated Thigh: Treatment with Trusculpt (Radio Frequency) Device
- Contra-lateral Untreated Thigh: No treatment with Trusculpt (Radio Frequency) Device
Arm/Group | Treated Thigh | Contra-lateral Untreated Thigh
Number analyzed (Participants) | 26 | 26
cm | .98 [-.30 to 2.05] | .32 [-.55 to 1.80]

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment
Groups:
- Untreated Thigh: No Treatment with RF device
Arm/Group | Treated Thigh | Untreated Thigh
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 41/44 | 0/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Thigh (N=44) | Untreated Thigh (N=44)
Erythema (Skin and subcutaneous tissue disorders) | 41 | 0
Edema (Skin and subcutaneous tissue disorders) | 13 | 0
Lumps (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No